CLINICAL TRIAL: NCT02234908
Title: Rewards for Tuberculosis Contact Screening
Acronym: RECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); City of Johannesburg (Unknown); Helen Joseph Hospital (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-33047; M140529 (Other: Wits University HREC (Medical)); 1U01AI100015-01 (NIH)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Tuberculosis; Drug-resistant Tuberculosis
Keywords: Tuberculosis; Drug-resistant tuberculosis; Incentives; Symptom screening
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contacts (Experimental): Contacts are the household contacts of confirmed TB and drug-resistant TB patients.
  Interventions: Behavioral: Contacts
- Index (Other): Index subjects are confirmed TB and drug-resistant TB patients who distribute referral cards to their household contacts.
  Interventions: Behavioral: Index

INTERVENTIONS:
Behavioral: Contacts — Household contacts who come to the study clinic, present a referral card, and complete TB symptom screening will receive a shopping voucher of $5-10 value.
  Arms: Contacts
Behavioral: Index — Index subjects will be entered in a prize lottery if any of their contacts complete TB symptom screening at the study clinic.
  Arms: Index

SUMMARY:
This pilot project is an evaluation of the feasibility, acceptability, and cost of offering an economic reward, in the form of a shopping voucher, to the household contacts of index patients (outpatient drug-susceptible and drug-resistant TB patients) who present at the study clinic for TB screening and optional HIV testing, providing a reward to the index patients for participating, and entering index patients whose contacts do present into a lottery to win a prize.The effectiveness of the intervention in screening a high proportion of contacts will be compared to existing published data from studies of active case-finding through home visits and of the status quo passive case finding. If successful, this pilot project will create a demand for screening among high risk patients, who will be rewarded for identifying themselves to the healthcare system, and could prove to be an affordable alternative to resource-intensive home visits. It will also shift responsibility for contact tracing from overburdened clinic staff to those who have the most to gain from early case detection-the patients and their families.

DETAILED DESCRIPTION:
Despite the success of antiretroviral treatment (ART) programs in reaching > 10 million HIV-infected patients in resource-limited countries over the past decade, HIV and tuberculosis (TB), continue to take a heavy toll on survival and health in southern Africa. In South Africa, where 6.4 million people are estimated to be HIV-positive and up to 2.1 million are on ART, TB incidence is the second highest in the world (after Swaziland), 65% of TB patients are HIV-infected, and TB remains the leading natural cause of death. Drug-resistant TB (DR-TB) is even more concerning, with more than 15,000 South African patients diagnosed with multidrug-resistant TB (MDR-TB) in 2012, nearly a fifth of the global total, and very high mortality among those receiving standard MDR-TB treatment.

Because of the high risk of both TB and HIV among the household contacts of TB patients and the importance of early case detection for both diseases and especially for DR-TB, improving TB case finding is a high priority. Recent studies have shown that having healthcare workers make multiple visits to the homes of TB patients in order to screen household contacts is a logistically challenging and resource- intensive strategy, and it is not routinely undertaken in most public sector settings in South Africa. One alternative to home visits that could prove effective and affordable is to offer small economic rewards to the household contacts of TB patients who voluntarily present at a healthcare facility for TB symptom screening and optional HIV testing. Economic incentives have been successful in increasing demand for healthcare in a variety of settings, but they have not been tried before as a way to increase uptake of services among patients' contacts, rather than among the diagnosed patients themselves.

This pilot project is an evaluation of the feasibility and results of offering an economic reward, in the form of a shopping voucher, to the household contacts of index patients (outpatient drug-susceptible and drug-resistant TB patients) who present at the study clinic for TB screening and optional HIV testing, providing a reward to the index patients for participating, and entering index patients whose contacts do present into a lottery to win a prize. The effectiveness of the intervention in screening a high proportion of contacts will be compared to existing published data from studies of active case-finding through home visits and of the status quo passive case finding. If successful, this pilot project will create a demand for screening among high risk patients, who will be rewarded for identifying themselves to the healthcare system, and could prove to be an affordable alternative to resource-intensive home visits. It will also shift responsibility for contact tracing from overburdened clinic staff to those who have the most to gain from early case detection-the patients and their families.

ELIGIBILITY:
Inclusion criteria for index cases:

* Adult patients (>18 years)
* Newly diagnosed with pulmonary TB (drug-susceptible or drug-resistant) or initiating treatment for TB at one of the study sites

Exclusion criteria for index cases:

* Resident outside the site's permissible catchment area for service delivery
* No household contacts (live alone)
* Admitted for inpatient care immediately following their TB diagnosis, and thus not readily able to distribute the referral cards
* Not physically, mentally, or emotionally able to participate in the study, in the view of study staff
* Previously enrolled in the same study
* Declines to provide written informed consent to participate
* Unable to speak any of the languages for which consent documents are available and not accompanied by person who can

Inclusion criteria for contacts:

* Usually spend at least 4 nights per week in the same household as an index case
* Can provide referral card given to contact by index patient

Exclusion criteria for contacts:

* Currently on any type of TB treatment
* Not able to present any form of identification that matches the information on the referral card
* Previously enrolled in the same study
* Declines to provide written informed consent to participate
* Unable to speak any of the languages for which consent documents are available and not accompanied by person who can

Inclusion criteria for interview respondents:

* Experience with the intervention as provider or patient
* Written informed consent to be interviewed

Exclusion criteria for contacts:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of household contacts volunteering for TB symptom screening | 30 days
  The primary quantitative outcome is uptake of TB symptom screening, defined as the proportion of reported household contacts who complete TB symptom screening within 1 month of index subject enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, Principal Investigator — Boston University
Locations (2):
- South Africa (2):
  - Helen Joseph Hospital, Johannesburg
  - OR Tambo Clinic, Johannesburg

IPD SHARING:
Plan to Share IPD: Undecided